CLINICAL TRIAL: NCT05454709
Title: A Stable Glucagon Analog Administered by a Bihormonal Closed Loop System; a Feasibility Study
Brief Title: A Stable Glucagon Analog Administered by a Bihormonal Closed Loop System
Acronym: STABLE-1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study medication could not be delivered by manufacturer.
Sponsor: Inreda Diabetic B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: NL76691.100.22
Record Dates: First submitted 2022-05-06; First posted 2022-07-12 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dasiglucagon; Glucagon-Like Peptide 1

STUDY DESIGN:
Intervention Model Description: Three days treatment A, four days wash out period (standard treatment), three days treatment B.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational Medicinal Product dasiglucagon and control GlucaGen are masked as either treatment A or B. Only the assistant researcher who does the preparation and allocation of the drugs has this key.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dasiglucagon (Experimental): Dasiglucagon 1mg/ml solution for subcutaneous injection. Size and frequency of dosing will be determined by the AP algorithm. Duration: 3 days.
  Interventions: Drug: Dasiglucagon
- GlucaGen (Active Comparator): Glucagon 1mg/ml solution for subcutaneous injection. Size and frequency of dosing will be determined by the AP algorithm. Duration: 3 days.
  Interventions: Drug: GlucaGen

INTERVENTIONS:
Drug: Dasiglucagon — Use of dasiglucagon in the AP system.
  Arms: Dasiglucagon
Drug: GlucaGen — Use of GlucaGen in the AP system.
  Arms: GlucaGen

SUMMARY:
The main objective is to determine the feasibility of dasiglucagon in a bi-hormonal reactive closed loop system for automated glucose regulation (artificial pancreas; AP®) in patients with diabetes mellitus type 1. Safety parameters and pharmacodynamics are compared between Dasiglucagon and GlucaGen®.

This study is a single-center, double-blinded, randomized, cross over trial in 12 subjects. The subjects will be randomized to receive either dasiglucagon or GlucaGen® for the first three day study period and switch to the alternate treatment after a wash-out treatment.

DETAILED DESCRIPTION:
Background of the study:

Inreda Diabetic B.V. (Goor, The Netherlands) developed a bi-hormonal reactive closed loop system to automate glucose regulation (artificial pancreas; AP) in patients with diabetes mellitus type 1. In the current CE-marked AP, GlucaGen® (Novo Nordisk, Denmark) is used as glucagon. This glucagon formulation is not stable and therefore fibrillation and infusion set occlusion could occur, resulting in reduced glucagon action with risk for hypoglycemia. Dasiglucagon (Zealand Pharma, Denmark) is a glucagon analog stable in aqueous solution and does therefore not suffer from fibrillation.

Objective of the study:

The main objective is to determine the feasibility of dasiglucagon in the Inreda AP-system. Secondary objectives are to assess safety parameters, differences in pharmacodynamics between dasiglucagon and GlucaGen® and differences in AP related outcomes.

Study design:

This study is a single-center, double-blinded, randomized, cross over trial which will be performed out-patient.

Study population:

The study population will comprise 12 subjects with diabetes type 1 using the AP system. Inclusion criteria are subjects from 18 years and older and treated with the Inreda AP system for a minimum of 1 month.

Intervention:

The intervention contains use of dasiglucagon administered by the Inreda AP-system. The subject will be randomized to receive either dasiglucagon or GlucaGen® during the first three days. After a wash-out period of four days, the subject will be switched to the alternate treatment. During both study periods subjects have to keep a diary, perform exercise, keep a WiFi access point with them, and have some eating restrictions.

Primary study parameters/outcome of the study:

Main parameter to express feasibility is the time in range (3.9 - 10.0 mmol/l), which will be compared between the dasiglucagon and reference glucagon.

Secondary study parameters/outcome of the study:

* Safety will be expressed as side effects of dasiglucagon compared to side effects of GlucaGen.
* The amount of extra food intakes to prevent/ combat hypoglycemia.
* Pharmacodynamics will be expressed in proportion of time spent in hypo-/hyperglycemia, median/mean glucose value, glycemic variability and PD curves, which will all be compared between the dasiglucagon and reference glucagon.
* AP related outcomes will be expressed in daily administered (maintenance) dosage of insulin/glucagon and the percentage of time that the closed loop algorithm is active.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes mellitus type 1;

  * Treated with the Inreda AP system for a minimum of 1 month;
  * Age between 18 and 75 years;
  * Adequate contraception is required (only applicable for female participants);
  * Willing and able to sign informed consent.

Since subjects are treated with the Inreda AP, the following inclusion criteria will be met:

* Treated with SAP or CSII for a minimum of 6 months;
* HbA1c < 97 mmol/mol;
* BMI < 35 kg/m2;
* No use of acetaminophen, as this may influence the sensor glucose measurements.

Exclusion Criteria:

* Impaired awareness of hypoglycemia (score ≥ 4) according to Gold and/or Clarke questionnaire [3], [4];

  * Pregnancy and/or breastfeeding;
  * Use of oral antidiabetic agents;
  * Pheochromocytoma;
  * Insulinoma;
  * Severe liver/heart/renal failure;
  * Alcohol abuse;
  * Hypersensitivity reactions to dasiglucagon, glucagon or any of the excipients;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-29 (Estimated); Primary Completion 2023-12-29 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Time in range | 3 days
  Time of glucose concentration in the range 3.9-10.0 mmol/L in %

SECONDARY OUTCOMES:
Side effects | 3 days
  Side effects of dasiglucagon and GlucaGen
Extra food intakes (food intake diary) | 3 days
  The participant is instructed to eat the same meals in the intervention and control period.
  Except extra food intakes when needed to prevent/combat hypoglycemia. Food intakes not present in the other period are extra food intakes.
Pharmacodynamics - hypo/hyper | 3 days
  Time spent in hypo-/hyperglycemia in percent
Pharmacodynamics - glucose value | 3 days
  Median glucose value in mmol/L
Pharmacodynamics - glycemic variability | 3 days
  Coefficient of variation (Standard deviation divided by the mean) in percent
Pharmacodynamics - glycemic variability | 3 days
  Inter quartile range in mmol/L
Pharmacodynamics - PD curves | 3 days
  Pharmacodynamics curves
AP related parameters - doses | 3 days
  Daily administered dose of insulin and glucagon in units
AP related parameters - algorithm | 3 days
  Time that algorithm is active in percent

CONTACTS AND LOCATIONS:
Overall Officials: G Laverman, MD, Principal Investigator — ZGT hospital
Locations (1):
- ZGT hospital, Almelo, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No